CLINICAL TRIAL: NCT02593669
Title: The Effect of Cataract Surgery for Age-related Cataract Patients on Circadian Rhythm and Sleep Quality
Brief Title: The Effect of Cataract Surgery on Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCPMOH2010-China8
Record Dates: First submitted 2015-10-28; First posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Cataract; Sleep
MeSH Terms: conditions — Cataract | interventions — Drug Implants; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neutral IOL (Experimental): Phacoemulsification cataract surgery is performed with neutral IOL implantation.
  Interventions: Procedure: Phacomulsification lens removal cataract surgery with neutral Intraocular lens(IOL) implantation; Drug: Subconjunctival dexamethasone and general anesthesia; Drug: Viscoelastic materials
- Blue-blocking IOL (Experimental): Phacoemulsification cataract surgery is performed with blue-blocking IOL implantation.
  Interventions: Procedure: Phacomulsification lens removal cataract surgery with blue-blocking Intraocular lens(IOL) implantation; Drug: Subconjunctival dexamethasone and general anesthesia; Drug: Viscoelastic materials

INTERVENTIONS:
Procedure: Phacomulsification lens removal cataract surgery with neutral Intraocular lens(IOL) implantation — The phacoemulsification lens removal cataract surgery is performed with neutral IOL.implantation
  Arms: Neutral IOL
Procedure: Phacomulsification lens removal cataract surgery with blue-blocking Intraocular lens(IOL) implantation — The phacoemulsification lens removal cataract surgery is performed with blue-blocking IOL.implantation.
  Arms: Blue-blocking IOL
Drug: Subconjunctival dexamethasone and general anesthesia — All patients received subconjunctival dexamethasone (2 mg) during surgery, and all surgeries were performed under general anesthesia.
Drug: Viscoelastic materials — viscoelastic materials are used to protect corneal endothelial cells.

SUMMARY:
A cataract is a clouding of the crystalline lens inside the eye, which leads to a decrease in vision. It is the most prevalent, treatable cause of visual impairment and blindness in the world. Cataract surgery with an intraocular lens (IOL) implant is one of the most common and thought to be the most effective surgical procedure in any field of medicine. In this trial, the investigators aimed to evaluate the effect of cataract surgery on circadian rhythm and sleep as well as the effect of the blue light transmission characteristics of the implanted IOL on sleep.

DETAILED DESCRIPTION:
A Prospective, randomized controlled study of 10000 participants(20000 eyes) with dense nucleus were enrolled. Patients were assigned to two groups: Group I: neutral IOL implanted in eye while in Group II, blue-blocking IOL was innovatively implanted in the eye.

A cataract is a clouding of the crystalline lens inside the eye, which leads to a decrease in vision. It is the most prevalent, treatable cause of visual impairment and blindness in the world. Cataract surgery with an intraocular lens (IOL) implant is one of the most common and thought to be the most effective surgical procedure in any field of medicine.

In this trial, the investigators aimed to evaluate the effect of cataract surgery on circadian rhythm and sleep as well as the effect of the blue light transmission characteristics of the implanted IOL on sleep. Patients enrolled into the study will be assessed in 3 months before the surgery and 3 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract scheduled for cataract surgery

Exclusion Criteria:

* Vision-impairing ophthalmic disease: Glaucoma, AMD, DR.et.al
* Severe systemic disease: Diabetes, Sleep disorder.et.al
* Vision-impairing complications: Ruptured posterior capsule, Persistent cornea edema.et.al

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from Post-illumination pupil response (PIPR) | 3 months before the surgery and 3 months after the surgery
Change from Objective sleep quality:actigraphy | 3 months before the surgery and 3 months after the surgery
Change from Subjective sleep quality: PSQI | 3 months before the surgery and 3 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D., Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Weirong Chen, M.D., Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Brondsted AE, Sander B, Haargaard B, Lund-Andersen H, Jennum P, Gammeltoft S, Kessel L. The Effect of Cataract Surgery on Circadian Photoentrainment: A Randomized Trial of Blue-Blocking versus Neutral Intraocular Lenses. Ophthalmology. 2015 Oct;122(10):2115-24. doi: 10.1016/j.ophtha.2015.06.033. Epub 2015 Jul 30. PMID 26233628
- [Background] Ayaki M, Negishi K, Tsubota K. Rejuvenation effects of cataract surgery with ultraviolet blocking intra-ocular lens on circadian rhythm and gait speed. Rejuvenation Res. 2014 Aug;17(4):359-65. doi: 10.1089/rej.2014.1550. PMID 24701992
- [Background] Ayaki M, Muramatsu M, Negishi K, Tsubota K. Improvements in sleep quality and gait speed after cataract surgery. Rejuvenation Res. 2013 Feb;16(1):35-42. doi: 10.1089/rej.2012.1369. PMID 23145881
- See also: Description Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/